CLINICAL TRIAL: NCT01510522
Title: Evaluate Adherence to Treatment With Glucophage Sachets Versus Tablets in Diabetes Type 2 Patients, Previously Treated With Metformin Tablets
Brief Title: Evaluate Adherence to Treatment With Glucophage Sachets Versus Tablets in Diabetes Type 2 Patients Previously Treated With Metformin Tablets
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200084-508; 2011-002508-34 (EudraCT Number)
Record Dates: First submitted 2011-12-30; First posted 2012-01-16 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes; Glucophage; Metformin; sachets; tablets
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucophage sachets (Experimental): Patients receive Glucophage sachets, the powder formulation for oral solution in sachets.
  Interventions: Drug: Glucophage
- Glucophage tablets (Active Comparator): Patients received Glucophage tablets.
  Interventions: Drug: Glucophage

INTERVENTIONS:
Drug: Glucophage — Glucophage Powder for oral solution in sachets (metformin hydrochloride in 850mg strengths) Dosing schedule: > 1.700mg/day for 6 month
  Other Names: Metformin hydrochloride
  Arms: Glucophage sachets
Drug: Glucophage — Glucophage tablets (metformin hydrochloride in 850mg strengths)
  Dosing schedule: > 1.700mg/day for 6 month
  Other Names: Metformin hydrochloride
  Arms: Glucophage tablets

SUMMARY:
This is an open-label, multicenter, two-arm, parallel, randomized phase 4 study to compare the compliance in diabetes type 2 patients treated with Glucophage sachets versus patients treated with Glucophage tablets.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 diagnosed (Baseline Glycemia > 7,0 mmol/L (126 mg/dL) or overload Glycemia > 11,0 mmol/L (198 mg/dL)
* On treatment with metformin tablets
* Patients with at least 2 treated co-morbidities
* Established dose of Metformin > 1.700 mg/day
* Age > 18 years old
* Given informed consent

Exclusion Criteria:

* Patients not able to take medication orally
* According to Summary of Product Characteristics (SmPC)
* Participating in another clinical trial 30 days prior to randomization
* Any other illness or medical or psychiatric condition, severe and uncontrolled that could interfere in the patient's participation or in the assessment of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Patient self-reported subjective compliance as assessed by Haynes-Sackett test at Month 6 | Month 6

SECONDARY OUTCOMES:
Objective compliance to treatment | Month 3 and month 6
  Objective compliance to treatment is assessed by the accountability of medication returned. Patient is assessed as compliant with an adherence of over 80%.
Evaluation of treatment satisfaction and preferences with the Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Baseline, month 3 and month 6
Rate of reported adverse events | Month 3 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck, S.L., Spain